CLINICAL TRIAL: NCT05621525
Title: A Phase I, Open Label, Dose Escalation and Expansion, Two- Part Study of SHP-2 Inhibitor BBP-398 to Evaluate the Safety, Tolerability, Pharmacokinetics and Preliminary Anti-cancer Activity in Chinese Subjects With Advanced Solid Tumors
Brief Title: Phase I Study of the BBP-398 in Patients With Advance Solid Tumors
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Business reason
Sponsor: LianBio LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LB1002-101
Record Dates: First submitted 2022-11-10; First posted 2022-11-18 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Advanced Solid Tumor; Advanced or Metastatic Non-small Cell Lung Cancer
Keywords: Solid Tumors, NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Part A Dose Escalation and Part B Dose Expansion (Experimental): Part A: Oral capsules taken in escalating levels to determine MTD/RP2D. Each treatment cycle will be 28 days in duration with BBP-398 administered, once daily (QD).
  Part B: Oral capsules administered at MTD/RP2D defined dose. Each treatment cycle will be 28 days in duration with BBP-398 administered, once daily (QD)
  Interventions: Drug: BBP-398

INTERVENTIONS:
Drug: BBP-398 — BBP-398 (formerly known as IACS-15509) is a potent, selective, orally active allosteric inhibitor of SHP2, a tyrosine phosphatase that plays a key role in the RTK -MAPK signal transduction pathway. Key components of the MAPK pathway include the small GTPase RAS, the serine/threonine-protein kinase RAF, mitogen-activated protein kinase (MEK) and ERK. In cells, SHP2 binds to phosphorylated tyrosine residues in the intracellular domain of RTKs such as the EGFR, leading to activation of the downstream MAPK signaling pathway.
  Other Names: IACS-15509

SUMMARY:
This is an open label, dose escalation and expansion, two-part Phase I study for SHP-2 inhibitor BBP-398 to evaluate the safety, tolerability, pharmacokinetics, determine MTD and/or RP2D, and preliminary anti- cancer activity in Chinese subjects with advanced solid tumors and in Chinese subjects with advanced or metastatic EGFR-mutant NSCLC.

DETAILED DESCRIPTION:
The Part A of this phase I trial is an abbreviated dose escalation study of BBP-398 following the USA mono dose escalation study (Study NAV- 1001, clinicaltrials.gov ID NCT04528836). The purpose of this part is to evaluate the safety, tolerability, pharmacokinetics, and preliminary anti-cancer activity in Chinese subjects with advanced solid tumors. The Part B of this study is to explore the safety, tolerability and efficacy of BBP-398 in Chinese subjects with advanced or metastatic EGFR- mutant NSCLC at MTD and/or RP2D. This Phase I study will provide supportive data to enable Chinese patients to join the combo dose escalation and expansion studies and/or other clinical trials of BBP-398.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have the ability to understand and the willingness to sign a written informed consent document 2 Patients must be willing and able to comply with the scheduled visits, treatment plan, laboratory tests and other specified study procedures 3. Age ≥18, male or female 4.Dose escalation: locally advanced or metastatic solid tumors Dose expansion: Advanced or metastatic EGFR-mutant NSCLC 5. Patients must have measurable disease by RECIST v1.1. 6. Patients must have an ECOG performance status (PS) ≤2 7.Patients with a life expectancy of ≥12 weeks. 8. Patients must have adequate organ function

Exclusion Criteria:

1. Patients with a known additional malignancy that is progressing or requires active treatment
2. Patients who have previously received a SHP-2 inhibitor
3. Patients who are hypersensitivity to SHP-2 inhibitor or any ingredients
4. Treatment with any of the related anti-cancer therapies prior to the first dose of BBP-398 within the stated timeframes
5. Patients with known active Hepatitis B, Hepatitis C infection, or HIV infection.
6. Patients with any of the cardiac-related issues or findings
7. Patients with a history of CVA, myocardial infarction or unstable angina within the previous 6 months before starting therapy.
8. Patients with known central nervous system (CNS) tumors
9. Patients with known active CNS metastases and/or carcinomatous meningitis.
10. Patients with persisting toxicity related to prior therapy.
11. Patients who have undergone major surgery within 4 weeks prior to study enrollment.
12. Pregnant or breastfeeding female patients.
13. Patients with inability to swallow oral medications or with gastrointestinal illness that would preclude the absorption of an oral agent.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2022-10-18 (Actual); Primary Completion 2024-03-29 (Actual); Study Completion 2024-03-29 (Actual)

PRIMARY OUTCOMES:
Determination of Maximum Tolerated Dose (MTD) of BBP-398 | Completion of 1 Cycle (28 days)
  The MTD will be based on DLT
Determination of anti-tumor activity of BBP-398 | Completion of 1 Cycle (28 days)
  Anti-tumor activity will be defined by objective response rate (ORR, complete response + partial response rate) and duration of response (DOR) according to RECIST v1.1

SECONDARY OUTCOMES:
Part A:Maximum plasma concentration (Cmax) of BBP-398 | Approximately 6 months
  Maximum plasma concentration of BBP-398 after single and multiple dose administration of BBP-398
Part A:Time to reach Cmax (Tmax) of BBP-398 | Approximately 6 months
  The amount of time to reach Cmax after single and multiple dose administration of BBP-398
Part A: Terminal half-life (t1/2) of BBP-398 | Approximately 6months
  Terminal half-life (t1/2) after single and multiple dose administration of BBP-398
Part A: Area under the plasma concentration-time curve (AUC) of BBP-398 | Approximately 6 months
  Area under the plasma concentration versus time curve after single and multiple dose administration of BBP-398
Part A: Concentration of BBP-398 in urine | Approximately 6 months
  To evaluate BBP-398 excretion via urine after single and multiple dose administration of BBP-398.
Part B: Concentration of BBP-398 in plasma | Approximately 6 months
  To evaluate BBP-398 plasma concentration after multiple dose administration of BBP-398.

CONTACTS AND LOCATIONS:
Overall Officials: Li Zhang, Master, Principal Investigator — West China Hospital; Yongsheng Wang, Doctor, Principal Investigator — West China Hospital
Locations (2):
- China (2):
  - Sun Yat-sen University Cancer Center, Guanzhou, Guangdong
  - West China Hospital Sichuan University, Chengdu, Sichuan